CLINICAL TRIAL: NCT00167063
Title: Falls in Stroke Patients After Hospital Discharge: Prevalence and Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 55m1
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Stroke
Keywords: Stroke; Fall; Fall prediction; Clinical manifestations; Frequent faller
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purposes of this study are: (1) to investigate the incidence and causes of falls of stroke patients residing in Taipei City and Taipei county after their discharge from the National Taiwan University Hospital, (2) to investigate the relationship between clinical manifestations of stroke patients before their hospital discharge and their incidence of falls after hospital discharge, and (3) to identify the risk factors for stroke patients who frequently fall after hospital discharge.

DETAILED DESCRIPTION:
Falls are one of the most common accidents among stroke patients. Stroke patients are more prone to falls than community-dwelling older adults because of their cumulative risk factors of falls such as cognitive impairment and motor dysfunction. Recent studies on falls in Taiwan have primarily focused on falls of community-dwelling older adults. Research focused on falls among stroke patients in Taiwan, however, is scarce. Studies reported by researchers in other countries have only investigated the incidence and causes of falls of patients staying in medical institutions up to three months post-stroke. Therefore, the incidence and immediate causes of falls remain unknown for post-hospital discharge stroke patients during their sub-acute and chronic stages. In addition, whether falls of stroke patients after hospital discharge could be predicted by their clinical manifestations during hospital stay also requires further investigation.

ELIGIBILITY:
Inclusion Criteria:

* between 40 and 75 years old
* first onset or recurrent stroke as a result of a single cerebral vascular accident (ischemic or hemorrhage stroke)
* ever received rehabilitation therapies at National Taiwan University Hospital
* being willing to take the clinical assessments
* residents of Taipei City or Taipei County

Exclusion Criteria:

* having unstable vital sign, unconsciousness, or having serious cognitive, perception, and language impairment, and being unable to follow the order of the experimenter
* having other neurological diseases(ex. Parkinson's disease or cerebellar disease etc.), or moderate to severe neuromuscular or musculoskeletal disorders, or disorders from systematic diseases those will influence the balance performance other than stroke

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-08; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Chein-Wei Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan